CLINICAL TRIAL: NCT04917380
Title: The Clinical Character，Risk and Prognosis of Post-neurosurgical Intracranial Infection With Different Pathogens.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0335
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Intracranial Infections; Ventriculitis; Meningitis; Gram-Positive Bacterial Infections; Gram-Negative Bacterial Infections; Neurosurgery
MeSH Terms: conditions — Meningitis; Gram-Positive Bacterial Infections; Gram-Negative Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gram-negative bacteria group: Gram-negative bacteria intracranial infection after neurosurgery
- Gram-positive bacteria group: Gram-positive bacteria intracranial infection after neurosurgery

INTERVENTIONS:
Other:  — Retrospective clinical study，no intervention

SUMMARY:
Intracranial infection is one of the common clinical complications after neurosurgery, especially after external cerebrospinal fluid drainage. Postoperative intracranial infection has a very high incidence, and its incidence is about 0.34%-3.1%. Once infection occurs, it will directly affect the length of hospitalization, mortality and disability of postoperative patients. The pathogenic bacteria of postoperative intracranial infections include G-bacteria and G+ bacteria, and fungi. Common G+ bacteria are Staphylococcus aureus. Common G-bacteria are Acinetobacter baumannii, Klebsiella pneumoniae, and Pseudomonas aeruginosa Bacteria, Escherichia coli and so on. In recent years, studies have reported that postoperative intracranial infections of G-bacteria are gradually increasing. In the previous study of our research group, it was found that Acinetobacter baumannii and Klebsiella pneumoniae accounted for the top two pathogens of postoperative intracranial infections in ICU. In particular, the proportion of carbapenem-resistant G-bacteria has increased, which brings difficulty and challenge to the treatment and seriously affects the prognosis of patients. Different pathogen infections may lead to different prognosis of patients with intracranial infection after neurosurgery. With different pathogens as the starting point, there are few studies comparing the clinical features, risk factors, and prognosis of intracranial infections after neurosurgery. Therefore, it is great significant to explore and understand different pathogenic bacteria, risk factors, drug resistance, treatment options, and prognosis after neurosurgery.

DETAILED DESCRIPTION:
1. To study the epidemiological distribution of pathogenic bacteria of intracranial infection after neurosurgery.
2. To study the risk factors of intracranial infection after neurosurgery (operations, type of external drainage tube, days of drainage tube , etc.).
3. To compare differences in clinical character，risks , treatment options, prognostic indicators between G+ bacterial infection group and G-infected bacterial group after neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with intracranial infection after surgery and positive pathogenic microorganisms cultured in cerebrospinal fluid

Exclusion Criteria:

* (1) < 18 years old, (2) Pregnant or lactating women, (3) fungus in CSF culture, (4) Clinical judgment is not intracranial infection, and CSF culture positive considers contaminating patients.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A retrospective review of the Second Affiliated Hospital of Zhejiang University from January 2013 to May 2021, diagnosed patients with intracranial infection after surgery and positive for pathogenic microorganisms cultured in cerebrospinal fluid.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-10 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 day mortality
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: 巍 崔, MD, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China